CLINICAL TRIAL: NCT03831659
Title: Prevalence of Migraine in Infertile Women and Evolution During in Vitro Fertilization (IVF)
Brief Title: Migraine and Infertility
Acronym: FERTIMIG
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180064
Record Dates: First submitted 2019-01-17; First posted 2019-02-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Migraine
Keywords: migraine; in vitro fertilization; infertility
MeSH Terms: conditions — Migraine Disorders; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: self-questionnaires — After collecting their non-opposition, a self-questionnaire will be given to them. This questionnaire is validated in the literature concerning the diagnosis of migraine. It includes questions about medical history and possible headaches

SUMMARY:
The purpose of this study is to determine the prevalence of migraine in infertile women and during in Vitro Fertilization protocol. Migraine is two to three times as common in women as in men. Migraine has considerable impact on quality of life. In Vitro Fertilization has become a common therapeutic modality in modern fertility medicines. Treatment protocols are associated with exaggerated hormonal fluctuations. Estrogen is considered to be closely linked to migraine and its fluctuations have been considered to trigger migrainous headaches.

DETAILED DESCRIPTION:
In Vitro Fertilization has become a common therapeutic modality in modern fertility medicines. Treatment protocols are associated with exaggerated hormonal fluctuations. Estrogen is considered to be closely linked to migraine and its fluctuations have been considered to trigger migrainous headaches.

Both migraine and infertility are associated with impaired quality of life.

Objectives: to assess the prevalence of migraine in infertile women and during in Vitro Fertilization protocol in order to improve the management of these patients.

Protocol:

Women coming to consult at the Port Royal infertility center and meeting the inclusion (infertile women without long-term analgesic treatment) criteria will be offered the study. The information note and no objection form will be given by the gynecologist receiving them for consultation. After collecting their non-opposition, a self-questionnaire will be given to them. This questionnaire is validated in the literature concerning the diagnosis of migraine. It includes questions about medical history and possible headaches. The patient fills it immediately and gives it to the investigator. As part of the usual management, and regardless of their answers to the questionnaire, some of the patients will be reviewed in consultation for the programming of an IVF. During this "incoming" consultation with one of the midwives of the unit, a schedule of migraine headaches will be given to the patients. They will keep it, will complete it in case of migraine, and will give it to the gynecologist during the embryo transfer or the doctor receiving the couple in consultation on day 7 in case of absence of embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* infertile women supported in reproductive medical assistance at the Port Royal infertility center
* aged between 18 and 40 years old

Exclusion Criteria:

* long-term analgesic treatment
* women under guardianship or curatorship

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Unit of assisted reproductive medicine in a University hospital
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
migraine | At inclusion
  Prevalence of migrainous in infertile women

SECONDARY OUTCOMES:
migraine | At 2 months
  Prevalence of migrainous in infertile women

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Port-Royal, Paris, France

IPD SHARING:
Plan to Share IPD: No